CLINICAL TRIAL: NCT05410665
Title: The Roles of IL-9/E-cadherin and Ferroptosis in Intestinal Mucosal Barrier Injury in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: YKK21134
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Sepsis; Intestinal Mucosal Barrier; Ferroptosis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis group: Adult septic patients admitted into the intensive care unit (ICU) of Nanjing First Hospital. The diagnostic criteria for sepsis were in accordance with the surviving sepsis guidelines.
  Interventions: Procedure: Standard treatments for sepsis
- Control group: Baseline data (including age, sex, body-mass index, disease severity scores) matched adult non-septic critical patients in our ICU.

INTERVENTIONS:
Procedure: Standard treatments for sepsis — Standard treatments for others
  Groups: Sepsis group

SUMMARY:
The investigators aim to evaluate the roles of IL-9/E-cadheirin and ferroptosis in the intestinal mucosal barrier injury of sepsis. The results of this study would lay the foundation for revealing the mechanisms of EEN improving immune imbalance of sepsis and provide a new idea to the early treatment of sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of sepsis
2. Within 3 days of sepsis onset before ICU admission
3. No artificial nutrition (enteral or parenteral nutrition) were provided before ICU admission

Exclusion Criteria:

1. Ileus
2. Digestive tract hemorrhage
3. Inflammatory bowel disease
4. Cancer or chronic organ dysfunction (e.g., hepatic or renal dysfunction)
5. Malnutrition or immunodeficiency
6. Long-term use of hormones

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic patients and baseline data (including age, sex, body-mass index, disease severity scores) matched adult non-septic critical patients in ICU.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of intestinal barrier injury incidence of intestinal barrier injury | 7 days
  intestinal barrier injury

SECONDARY OUTCOMES:
Incidence of ferroptosis | 7 days
  ferroptosis

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kui Sun, Dr., Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided